CLINICAL TRIAL: NCT00005503
Title: Epidemiology of Cardiac Development in Youth
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5021; R03HL059223 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To document normal developmental changes in cardiac structure and function during late childhood and adolescence.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The investigators documented the nature and extent of changes in cardiac structure based on M-mode measurements and developed corresponding reference values. They documented the nature and extent of changes in cardiac function based on pulse Doppler measures and indices and developed corresponding reference values. They also investigated clinical findings based on M-mode and Doppler measurements as well as changes in body size and composition, sexual maturation, and other covariates. They used existing data from Project HeartBeat! 's 12 four-monthly examinations over the age range from 8 to 17 years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1997-09; Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darwin Labarthe — University of Texas